CLINICAL TRIAL: NCT06115057
Title: The Investigation of Gastrointestinal Tolerance of a Novel Fibre Blend Among ≥45-<70-year-old Men and Women
Brief Title: Fiber Tolerance Study
Acronym: Gitomix
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nutricia Research (Industry)
Collaborators: NCRU (Nutrition Clinical Research Unit) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23REX0058665; NL84292.056.23 (Other: CCMO, The Netherlands)
Record Dates: First submitted 2023-09-18; First posted 2023-11-02 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Tolerance of Dietary Fiber
Keywords: Fiber Tolerance Gastro-intestinal Safety
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Intervention Model Description: open-label, single-arm, single-site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Fiber
  Interventions: Dietary Supplement: Fiber

INTERVENTIONS:
Dietary Supplement: Fiber — Subjects in this study are to consume the study product twice daily during regular meals.
  The fiber mix consists of different types of dietary fiber that are individually well tolerated for human consumption.

SUMMARY:
Research shows that many people do not get enough dietary fiber through their normal diet. As a result, some nutrients are not properly absorbed into the bloodstream. The immune system however does need these nutrients. Dietary fibers are therefore important for health. Nutricia has developed a new blend of natural fibers that can help people get enough fiber.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 45 and ≤ 70 years
2. Body Mass Index (BMI) ≥ 18.5 and ≤ 29.9 kg/m2
3. Signed consent form
4. Willingness and ability to comply with the protocol
5. Good general health
6. Defecation frequency: between three bowel movements per week and three bowel movements per day within a month for screening.

Exclusion Criteria:

1. Presence or history of chronic gastrointestinal disorders (e.g. stomach ulcers, ulcerative colitis, Crohn's disease) or history of abdominal surgery with resection of the bowel (small or large intestine).
2. Presence of other medical conditions where gastrointestinal function often/probably is affected, such as:

   1. autoimmune diseases (e.g. diabetes mellitus type I, multiple sclerosis, systemic lupus erythematosus).
   2. eating disorders (e.g. anorexia nervosa, bulimia nervosa, binge eating disorder).
   3. intestinal/gastrointestinal disorder due to a stroke.
3. Chronic diseases (including but not limited to hypertension, dyslipidaemia, type 2 diabetes mellitus, thyroid disorders) that cannot be controlled with the use of medication/therapy.
4. Severe acute liver disease or chronic liver disease.
5. Severe or chronic kidney disease or need for hemodialysis.
6. Colonoscopy, irrigoscopy or other bowel cleansing, or other surgical procedures related to the gastrointestinal tract (eg. colon polypectomy, appendectomy) or for which use of systemic antibiotics within 1 month before the screening is required or scheduled during participation in the study.
7. Use of enemas, laxatives, antacids, proton pump inhibitors, prokinetics (e.g. metoclopramide, drugs that affect motility), digestive enzymes, narcotic/morphine analgesics within 1 week prior to screening or intended use during participation in the study.
8. Following a vegetarian or vegan diet.

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
GSRS change | 4 weeks
  Change from baseline in the reported severity of GI symptoms assessed by the Gastrointestinal Symptom Rating Scale (GSRS) for diarrhea dimension at week 4 post-baseline.

SECONDARY OUTCOMES:
GSRS change | week 1, week 2, week 3,
  Weekly changes from baseline in the reported severity of GI symptoms assessed by the GSRS for diarrhea dimension at week 1, week 2, and week 3 post-baseline.
GSRS change | week 1, week 2, week 3, week 4
  Weekly changes from baseline in the reported severity of GI symptoms assessed by the GSRS for abdominal pain, constipation, indigestion, and reflux dimensions at week 1, week 2, week 3, and week 4.

OTHER OUTCOMES:
GSRS | week 1, week 2, week 3, week 4
  The reported severity of GI symptoms assessed by the GSRS between week 1 v week 2, week 1 v week 3, week 1 v week 4, week 2 v week 3, week 2 v week 4, and week 3 v week 4 [score].
BSFC | week 1, week 4
  Weekly average faecal form type assessed by the Bristol Stool Form Chart at each defecation in the baseline week, at week 1, and week 4 post-baseline.
Defecation frequency | week 1, week 2, week 3, week 4
  Weekly average frequency of defecation, derived from the number of faecal form types assessed by the Bristol Stool Form Chart.
DQLQ | 4 weeks
  Digestion-associated Quality of life assessed by the Digestion-associated Quality of Life Questionnaire (DQLQ) at baseline and at week 4 post-baseline.
Stool | week 2, week 3, week 4
  Microbiota and other outcome parameters assessed using collected faecal samples in the baseline week and every 7 days over 4 weeks post-baseline:
  * Composition, diversity, and abundance of microbiota using 16S rRNA gene sequencing and processing
  * Short-chain fatty acids (SCFA)
  * Branch-chain fatty acids (BCFA)
  * Lactate
  * Ammonia
  * Calprotectin
  * Secretory immunoglobulin A (sIgA)
  * pH

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition Clinical Research Unit, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No